CLINICAL TRIAL: NCT00083096
Title: Phase I Study Of SCH66336 (Lonafarnib), A Farnesyl Protein Transferase Inhibitor In Combination With Temozolomide In Gliomas
Brief Title: Lonafarnib and Temozolomide in Treating Patients With Recurrent Primary Supratentorial Gliomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-16027-26023; EORTC-16027; EORTC-26023; SPRI-P03174
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult mixed glioma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult pilocytic astrocytoma; adult anaplastic ependymoma; adult subependymoma; adult myxopapillary ependymoma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult diffuse astrocytoma; adult subependymal giant cell astrocytoma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma; Ependymoma; Glioma, Subependymal; Gliosarcoma | interventions — lonafarnib; Temozolomide

INTERVENTIONS:
Drug: lonafarnib
Drug: temozolomide

SUMMARY:
RATIONALE: Lonafarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving lonafarnib together with temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lonafarnib when given together with temozolomide in treating patients with recurrent primary supratentorial glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxicity of lonafarnib when administered with temozolomide in patients with recurrent primary supratentorial gliomas.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Determine the mechanism of action of lonafarnib in these patients.
* Determine the pharmacodynamics and pharmacokinetics of this regimen in these patients.
* Determine the activity of this regimen in these patients.
* Determine the response to this regimen in patients who have measurable disease.

OUTLINE: This is a nonrandomized, multicenter, open-label, dose-escalation study of lonafarnib.

Patients receive oral temozolomide once daily on days 2-6 of course 1 and on days 1-5 of all subsequent courses. Patients also receive oral lonafarnib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of lonafarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 1 of 6 patients experience dose-limiting toxicity. An additional 3 patients may be treated at the highest dose level achieved.

Patients are followed every 8 weeks for 6 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary supratentorial glioma

  * Multifocal disease allowed
* Recurrent disease after prior surgery and/or radiotherapy
* Radiological evidence of increased and/or enhanced target lesion
* Amenable to temozolomide therapy

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2 OR
* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL

Hepatic

* Alkaline phosphatase < 2.5 times upper limit of normal (ULN)
* Transaminases < 2.5 times ULN
* Bilirubin < 1.5 times ULN

Renal

* Creatinine < 1.7 mg/dL

Cardiovascular

* Cardiac function clinically normal
* Normal 12-lead ECG
* QTc ≤ 440 msec on ECG
* No ischemic heart disease within the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No unstable systemic disease
* No active uncontrolled infection
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up
* No other active or recurrent malignancy within the past 5 years except cone biopsied carcinoma of the cervix or adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer biologic agents

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for temozolomide)
* Prior adjuvant chemotherapy allowed
* No more than 1 prior chemotherapy regimen for recurrent disease
* No other concurrent chemotherapy

Endocrine therapy

* Concurrent corticosteroids allowed provided treatment remains at a stable or decreasing dose for at least 2 weeks

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 3 months since prior surgery for primary brain tumor

Other

* Concurrent anticonvulsants allowed
* No other concurrent anticancer agents
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-03; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose of lonafarnib determined by CTCAE v3.0

SECONDARY OUTCOMES:
Response (complete [CR] or partial response [PR]) measured by McDonald's criteria at least 4 weeks after first documented response and every 8 weeks until disease progression or until start of another treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mario Campone, MD, Study Chair — Centre Regional Rene Gauducheau
Locations (3):
- France (2):
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland